CLINICAL TRIAL: NCT05517655
Title: BEGIN Novel ImagiNG Biomarkers
Acronym: BEGINNING
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of Kansas (Other); University of Iowa (Other); University of Virginia (Other)
Responsible Party: Principal Investigator, Jason Woods, Principal Investigator, Children's Hospital Medical Center, Cincinnati
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2021-0325
Record Dates: First submitted 2022-04-06; First posted 2022-08-26 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pre Trikafta (Experimental): 129Xe MRI
  Interventions: Drug: 129Xe
- Post Trikafta (Experimental): 129Xe MRI
  Interventions: Drug: 129Xe

INTERVENTIONS:
Drug: 129Xe — Rapid spatial mapping of lung, liver, and pancreatic structure and function is now possible with a combination of hyperpolarized 129Xe and traditional proton MRI, all absent sedation and ionizing radiation.

SUMMARY:
To determine the treatment effect of triple-combination therapy in 6-8 year olds after presumed FDA approval, using rapid structural and functional pulmonary and abdominal MRI (UTE and 129Xe).

DETAILED DESCRIPTION:
The overall hypothesis is that multi-organ MRI will provide more sensitive, robust outcome measures in young CF patients than traditional measures employed in the BEGIN study and that these novel measures will be more sensitive to treatment effects, tested here by comparison before and after triple-combination modulator therapy. By understanding the nature of early lung obstruction and characteristic changes in the liver and pancreas over time, we continue to lay the groundwork for more personalized medicine in the future.

Assessing treatment response and clinical benefit in children with CF who are clinically normal per standard outcomes (e.g., spirometry, pancreatic function) will become paramount as triplecombination therapy is extended to younger patients with milder CF clinical presentation than their historic peers. Here the sensitivity and profile free of ionizing-radiation exposure of MRI can be leveraged to follow an individual with CF over time to quantify changes with therapy-with additional spatial resolution unavailable from standard clinical testing.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (and assent where appropriate) obtained from the subject or subject's legal representative.
2. Willingness to adhere to the study-visit schedule and other protocol requirements.
3. Ages 6-8 years old at baseline MRI visit (may be enrolled up to 60 days before 6th birthday).
4. Documentation of CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype and one or more of the following criteria:

   1. Sweat chloride equal to or greater than 60 mEq/liter by quantitative pilocarpine iontophoresis test
   2. Two well-characterized mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene
5. Physician intent to prescribe triple-combination therapy
6. Clinically-stable with no respiratory tract infection at the time of enrollment.
7. No change in chronic maintenance therapies in the 28 days prior to enrollment.
8. Ability to cooperate with MRI procedures

Exclusion Criteria:

1. Individuals currently on ivacaftor therapy (including Kalydeco, Orkambi, and Symdeko) and with at least one gating mutation. Gating mutations include G551D, G178R, S549N, S549R, G551S, G970R, G1244E, S1251N, S1255P, or G1349D.
2. Acute respiratory symptoms (e.g. wheezing) at the time of the MRI.
3. Acute respiratory infection, defined as increased cough, wheezing or respiratory rate in the 28 days prior to enrollment.
4. Chronic lung disease not related to CF
5. Chronic liver disease not related to CF
6. Acute pancreatitis, defined by clinical criteria (45).
7. Chronic pancreatic disease not related to CF.
8. Physical findings that would compromise the safety of the subject or the quality of the study data as determined at the discretion of the site investigator.
9. Any other condition that, in the opinion of the Site Investigator/designee, would preclude informed consent or assent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Ventilation Defect Percentage change from baseline | 1 year
  For pulmonary MRI, the primary outcome measure is the change in 129Xe ventilation defect percentage (VDP) from pre-therapy baseline to the one-year follow-up visit.
Pancreas volume | 1 year
  For pancreatic MRI, the primary outcome measure is change in pancreas volume normalized to BSA between pre-therapy baseline and one-year follow-up visit.

SECONDARY OUTCOMES:
Abdominal T1 values | 1 year
  Changes in MRI T1 average in the liver and pancreas, from baseline to follow up at 1 year
Lung reader score | 1 year
  Changes in reader score for visible structural defects from proton MRI, from baseline to follow up at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jason Woods, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (3):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Carrie Stevens, Cincinnati, Ohio
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided